CLINICAL TRIAL: NCT01244321
Title: A Controlled, Single-Center Clinical Pilot Study to Evaluate the Performance of CoSeal as a Barrier for Adhesion Prevention in Patients Submitted to Ventricular Assist Device VAD)
Brief Title: COVADIS Pilot Trial: COseal in Ventricular Assist DevIceS
Acronym: COVADIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: COVADIS002
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: End-stage Heart Failure Awaiting VAD Implantation
Keywords: End stage heart failure; heart transplantation; Ventricular assist device; Patients with end stage heart failure; awaiting heart transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CoSeal Group: Subjects with indication for LVAD implantation, meeting the requirements for LVAD implantation. Patients for whom LVAD removal is anticipated not earlier than 6 weeks after LVAD implantation.
- CoSeal Control Group: Subjects who had a LVAD for more than 6 weeks.

SUMMARY:
The objective of this controlled, non-randomized, single-center pilot study (CoSeal arm prospective)study is to evaluate the efficacy of the synthetic surgical hydrogel CoSeal® in the prevention of cardiac adhesion formation in patients submitted to VAD procedures.

DETAILED DESCRIPTION:
In the past decade the use of ventricular assist devices) (VADs) for bridging to heart transplantation (HTx) or, in some cases, to recovery of the ventricular function has increased and, during the same time, the duration of the implantation period has lengthened dramatically. When removing VADs after a long period, surgeons face severe pericardial adhesions at the mediastinum level and of the surrounding tissue due to the inflammatory response. During resternotomy, dissection of these adhesions increases surgical time and can be a source of lesions on the cardiac or vascular structures and of severe bleeding at the moment of transplantation or when the device is removed.

Many products have been used to prevent or reduce adhesions but an ideal antiadhesive treatment has remained elusive. CoSeal®, a licensed synthetic hydrogel (Baxter, USA) has been shown to reduce pericardial adhesions in a limited series of reoperations.

ELIGIBILITY:
Inclusion criteria (CoSeal group):

1. Written informed consent obtained from the subject prior to participation in the study
2. At least 18 years of age
3. Subjects with indication for LVAD implantation, meeting the requirements for LVAD implantation. Patients for whom the investigator anticipates LVAD removal not earlier than 6 weeks after LVAD implantation.

Inclusion criteria (CoSeal control group):

1. Written informed consent obtained from the subject prior to participation in the study
2. At least 18 years of age
3. Subjects who had a LVAD for more than 6 weeks.

Exclusion criteria (CoSeal group):

1. Concomitant use of any other anti-adhesion product
2. Immune system disorders, immuno-deficiencies or immuno-suppression
3. Known hypersensitivity to components of the study product
4. Patients concurrently participating in another clinical trial for adhesion prevention or sealing evaluation and having received such an investigational drug or device within the previous 30 days
5. Patients who were previously subject to another LVAD implantation/explantation
6. Pregnant or breast-feeding women.

Exclusion criteria (Co Seal control group):

1. Known use of any other anti-adhesion product during VAD implantation
2. Immune system disorders, immuno-deficiencies or immuno-suppression
3. Patients concurrently participating in another clinical trial for adhesion prevention or sealing evaluation and having received such an investigational drug or device within the previous 30 days
4. Patients who were previously subject to another LVAD implantation/explantation
5. Pregnant or breast-feeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage heart failure, awaiting heart transplantion, with need for VAD (ventricular assist device)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Presence and severity of adhesions | At the moment of VAD-Removal/Transplantation (>6 weeks after VAD implantation)
  Assessment of adhesions using a scoring system, assessing six different sites.

SECONDARY OUTCOMES:
Bleeding | At the moment of VAD-Removal/Transplantation
  Hemostasis time (START: off pump time; STOP: skin closure); bleeding volume Tansfusions of blood related products - defined as quantity of blood related product transfusions (ml) administered to the patient from skin incision to discharge or 30 days after surgery, whichever comes first, for both first and second study operation Blood loss in chest drains - defined as amount of blood lost in the chest drains from postoperative time to discharge or 30 days after surgery, whichever comes first.
Clinical outcome | At the moment of VAD removal/transplantation (>6 weeks after VAD implantation)
  Surgery times (duration) during explantation/transplantation
  1. Dissection time (START: skin incision; STOP: on-pump time)
  2. Dissection time by region dissected, calculated as time to go to bypass (START: skin incision; STOP: initiation of bypass) by number of the investigational regions with adhesions dissected in this interval
  3. Time to VAD removal (START: skin incision; STOP: time of VAD removal from patient's chest at 2nd study operation)
  4. Length of operation (START: skin incision; STOP: chest closure).
Adhesion related | At the moment of VAD-Removal/Transplantation (>6 weeks after VAD implantation)
  1. Percentage of patients with grade 3 adhesions at VAD grafts
  2. Mean incidence score
  3. Mean adhesion severity score
  4. Percentage of sites free of adhesions
  5. Time required for adhesion dissection - pure dissection time before and after the CPB

CONTACTS AND LOCATIONS:
Overall Officials: Roland Hetzer, MD, PhD, Principal Investigator — Deutsches Herzzentrum Berlin, Germany
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany

REFERENCES:
- See also: Homepage of Deutsches Herzzentrum Berlin — http://www.dhzb.de